CLINICAL TRIAL: NCT03621319
Title: Eradicating Barrett's Esophagus Using Radiofrequency Ablation or a Novel Hybrid Argon Plasma Coagulation Technique (BURN)
Brief Title: Eradicating Barrett's Esophagus Using Radiofrequency Ablation or a Novel Hybrid Argon Plasma Coagulation Technique
Acronym: BURN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closure due to the COVID-19 pandemic: Protocol specified procedures could not be followed resulting in unavoidable protocol deviations. Lower enrollment than expected. Competing COVID-19 studies at study sites. No ethical, scientific, safety issues.
Sponsor: Erbe Elektromedizin GmbH (Industry)
Collaborators: Erbe USA Incorporated (Other); Kansas City Veteran Affairs Medical Center (U.S. Federal Agency); NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015_1
Record Dates: First submitted 2018-07-19; First posted 2018-08-08 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Barrett's Esophagus; High-grade Dysplasia in Barrett Esophagus; Low Grade Dysplasia in Barrett Esophagus
Keywords: Hybrid argon plasma coagulation; Submucosal injection
MeSH Terms: conditions — Barrett Esophagus | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Hybrid argon plasma ablation (HAPC) (Active Comparator): Eligible participants will be randomized to receive ablation of dysplasia with Hybrid argon plasma coagulation (HAPC) after EMR of visible lesions (if present) has been performed as per standard of care.
  Interventions: Device: Hybrid argon plasma ablation (HAPC)
- Radiofrequency ablation (RFA) (Active Comparator): Eligible participants will be randomized to receive treatment of dysplasia with RFA after EMR of visible lesions (if present) has been performed as per standard of care.
  Interventions: Device: Radiofrequency ablation (RFA)

INTERVENTIONS:
Device: Hybrid argon plasma ablation (HAPC) — -The assigned HAPC ablation will be performed at 8 to 12 week intervals until eradication of BE has been achieved or a total of 4 treatments have been performed
  Arms: Hybrid argon plasma ablation (HAPC)
Device: Radiofrequency ablation (RFA) — -The assigned RFA procedure will be performed at 8 to 12 week intervals until eradication of BE has been achieved or a total of 4 treatments have been performed
  Arms: Radiofrequency ablation (RFA)

SUMMARY:
Lay summary: Barrett's Esophagus (BE) involves a change of the esophagus lining (BE epithelium) which in a small proportion of patients could be the starting point for the development of cancer (esophageal adenocarcinoma). Currently, there is evidence that this change is initiated by acid reflux from the stomach which then could progress in a stepwise manner from the healthy epithelium to cellular changes (intestinal metaplasia, low-grade and high-grade dysplasia) and finally to adenocarcinoma. Surgery is considered the standard therapy for this cancer which involves the risk of death and complications with quality of life impairments. New possibilities for treatment have evolved with endoscopic therapies which allow for treatment of early changes of the epithelium (intestinal metaplasia and dysplasia) prior to the occurrence of cancer using either argon plasma coagulation (APC) or radiofrequency ablation (RFA). Both are established methods for eradication of BE by thermal ablation of the BE epithelium using high frequency current (HF). More advanced BE epithelium with early visible cancers are being treated by endoscopic mucosal resection (EMR). After EMR the residual Barrett's epithelium can also be removed by ablation with RFA or APC. Currently radiofrequency ablation (RFA) has been suggested as the standard therapy for BE treatment. Although effective in the eradication of the BE epithelium after RFA treatment the re-appearance of BE epithelium and the occurrence of complications such as strictures causing swallowing impairments for food have also been observed in clinical studies. A recently developed method is Hybrid argon plasma coagulation (ablation) [HybridAPC® (HAPC)] which combines argon plasma coagulation (APC) with a fluid injection function by a water beam. The water beam allows to establish a fluid cushion (normal sterile saline) right beneath the BE-epithelium prior to thermal ablation thereby protecting the esophagus wall from heat during ablation of epithelium with APC. The goal of this randomized controlled study is to investigate if HAPC is non-inferior to RFA in the stricture-free eradication of the dysplastic BE epithelium.

DETAILED DESCRIPTION:
Barrett's Esophagus (BE) is a pre-malignant condition and may progress to low grade dysplasia, high grade dysplasia and ultimately esophageal adenocarcinoma which has poor prognosis with a 5-year survival rate of only 5 - 20 %. Radiofrequency ablation (RFA) is a standard modality and well-studied endoscopic treatment for dysplastic BE. HybridAPC® (HAPC) is a newer technique for endoscopic treatment of dysplastic BE that involves submucosal fluid injection prior to performing APC. The study aim of this non-inferiority study is to show that HAPC is at least as safe and effective as RFA in the stricture-free eradication of dysplasia (CE-D).

The study is a multi-center, parallel group (HAPC/RFA) prospective, single blind, non-inferiority, randomized controlled study to assess the safety and effectiveness of HAPC (treatment arm) compared to RFA (control arm) in the treatment of BE in up to 144 male and female adult patients. Participants of the study will be enrolled in up to 15 centers in the US. Both techniques have never been directly compared in the treatment of BE.

The specific aim of this non-inferiority study is to show that HAPC is at least as safe and effective as RFA in the stricture-free eradication of dysplasia (CE-D), by inducing complete eradication of dysplasia (CE-D) within 12 months after last treatment as confirmed by endoscopy and histology.

HybridAPC® is an endoscopic technique that is used with the HybridAPC® Probe, the Water Jet Model ERBEJET 2 and an ERBE Argon Plasma Coagulator (APC) Model APC 2/Electrosurgical Unit (ESU) VIO Model System. The Water Jet delivers pressurized sterile 0.9 % sodium chloride solution (normal saline) through the HybridAPC® Probe into the submucosa of the Barrett mucosa. Reduction/limitation of unwanted tissue damage (penetration depth) is being ensured by the saline cushion when applying argon plasma coagulation to ablate Barrett's mucosa with subsequent regeneration of esophageal squamous mucosa.

Radiofrequency ablation (RFA) applied in the control arm using BarrxTM FLEX RFA Generator is an endoscopic technique that delivers high radiofrequency waves using either circumferential (balloon inserted over an endoscopically placed guidewire) device of focal (probe attached to the tip of the endoscope) device to damage the Barrett's mucosa with subsequent regeneration of esophageal squamous mucosa. While a circumferential device can be used to treat larger BE areas, focal device (Halo 60, 90 or through the scope device) can be used to treat small islands of residual BE. The depth of the injury is controlled by regular spacing of the electrodes and the delivery of a pre-set amount of energy through the probes. The PI/Co-investigators will be instructed to operate the BarrxTM FLEX RFA Generator and above referenced catheters according to the cleared labeling.

Patients with dysplastic BE will be identified at each participating center, and defined as those with LGD within previous 6 months and HGD/cancer within previous 6 months, both timed from date of consent. All histology slides from biopsies and endoscopic mucosal resection (EMR) specimens will be read by the local pathologist for patient management purposes and separately by a single independent reference pathologist to confirm patient eligibility for randomization.

Eligible patients will be block randomized at each participating study center at a ratio of 1 : 1 to receive treatment of dysplasia with HAPC or RFA after EMR of visible lesions (if present) has been performed as per standard of care. All patients will be assigned a unique registration number allocated by the Electronic Data Capture (EDC) system following details submitted on a web form. Due to the nature of the intervention only the patient will be blinded (single blinding), and not the PI or Co-investigators. The assigned HAPC ablation or RFA procedure will be performed at 8 to 12-week intervals until eradication of BE has been achieved. A maximum number of 4 treatment sessions is allowed.

Once the BE has been eradicated endoscopically, 4 quadrant biopsies every 1-2 cm will be performed to confirm complete eradication of dysplasia/IM (standard of care) and slides sent for confirmation by the central pathologist.

Primary statistical analysis will compare the proportions of patients in whom stricture-free eradication of dysplastic BE has been achieved.

As secondary endpoints complete endoscopic and histological eradication of intestinal metaplasia (CE-IM), stricture rate, post-operative pain, cost-effectiveness and recurrence of intestinal metaplasia and dysplasia will be documented and reported. No formal tests of hypothesis will be applied for these secondary endpoints.

Data from the trial will be entered into a database (VISION EDC, version 8, Prelude Dynamics, Austin, TX) and all statistical analyses will be performed using validated software (SAS, version 9.4; IBM/SPSS, version 23; Cytel StatXact, version 11; or R).

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-85 years (inclusive)
* Dysplastic BE, confirmed by the central pathologist; specifically:

  * Low grade dysplasia documented on biopsy within 6 months of consent date or
  * High grade dysplasia documented on biopsy within 6 months of consent date
* Barrett's extent of: C/M≥1 cm and C/M ≤ 6 cm using the Prague criteria [C = circumferential extent of disease / M = maximum extent of disease]
* Ability to provide written and informed consent

Exclusion Criteria:

* Barrett's extent of: C/M <1 cm or a C/M-value > 6 cm using the Prague criteria
* Prior EMR (endoscopic mucosal resection) for G3/G4; L1; V1; R1 (vertical margin only) or submucosal invasion;
* Presence of endoscopically visible abnormalities at the time of initial study treatment with HAPC or RFA. These participants can undergo EMR and then continue in the trial after a suitable healing period, provided randomization can occur within 90 days of consent.
* Presence of invasive cancer on biopsy
* Known pregnancy or plans to become pregnant
* Complete eradication is not considered a relevant treatment goal or in whom additional treatment is contraindicated;
* pre-existing significant esophageal pain or dysphagia;
* BE >80% has been resected by EMR;
* incomplete wound healing 3 months post-EMR despite adequate PPImedication;
* Prior ablative therapy in the esophagus but prior EMR allowed
* Active esophagitis or stricture precluding passage of scope
* Presence of esophageal varices
* Anticoagulant therapy (apart from aspirin or NSAIDS) that cannot be discontinued prior to therapy or uncorrectable hemostatic disorders
* Life expectancy less than 2 years
* Previous gastrectomy or other gastric surgery other than uncomplicated fundoplication

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Rate of stricture-free eradication of dysplastic BE | 12 months
  Freedom from strictures and complete eradication of dysplasia (CE-D) within 12 months after the last treatment will be measured as a composite safety and effectiveness endpoint. The composite endpoint evaluation is a traditional responder analysis with a single measure. The composite endpoint will have two possible outcome responses for each study subject: success or failure. The study or control treatment will be considered a success for a study subject only if both conditions are met: freedom from strictures and complete eradication of dysplasia. The number of successes and failures allows the estimation of success rates in the two study arms. These rates will be compared using standard statistical methods for rates (that is, binomial proportions).

SECONDARY OUTCOMES:
Rate of eradication of intestinal metaplasia (CE-IM) | 12 months
  Eradication of intestinal metaplasia (CE-IM) within 12 months after the last treatment will be measured
Post-operative pain | 7 days
  Post-operative pain score at baseline and at 1st and 7th day visits post treatment utilizing a visual analog scale (VAS). The VAS scale consists of a straight line with the scale endpoints defining extreme limits such as 'no pain' at "0" up to 'worst possible pain' at "10". The higher the value in the scale, the higher the pain intensity. A continuous 10 cm interval on which a subject marks a position is turned into a measurement (usually a fractional value like 5.5 cm). A lower value is thus a better outcome whereas a higher number indicates a worse outcome, with respect to pain intensity.
Major complications | 12 months
  Complications requiring additional Intervention (bleeding with drop of hemoglobin (Hb > 2 g/dl), fever persisting more than 24 hours, stricture, perforation)
Minor complications | 12 months
  Complications without need for additional endotherapy (bleeding with drop in hemoglobin (Hb < 2 g/dl) fever persisting less than 24 hours, dysphagia)
Recurrence rate of dysplasia (CE-D) | 12 months
  The recurrence rate of dysplasia after CE-D has been achieved will be measured
Recurrence rate of intestinal metaplasia (CE-IM) | 12 months
  The recurrence rate of intestinal metaplasia after CE-IM has been achieved will be measured
Cost-effectiveness of HAPC vs. RFA in the treatment of dysplastic BE | 12 months
  The cost effectiveness of HAPC compared to RFA for achieving CE-D will be based on a comparison of average treatment cost between the two groups. Data regarding the type of off-study medical services utilized during the study period that are possibly or definitely related to the ablative treatment will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Kansas City Veterans Affairs Medical
Locations (13):
- United States (13):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California, Irvine, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Veterans Affairs Hospital, Kansas City, Missouri
  - Washington University, School of Medicine; Department of Internal Medicine; Division of Gastroenterology, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center; Division of Digestive and Liver Diseases, New York, New York
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Utah School of Medicine, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No